CLINICAL TRIAL: NCT04908163
Title: Feasibility Study for the Development of a Nutritional-culinary Programme to Tackle Overweight or Obesity as a Strategy to Promote Adherence to a Healthy Dietary Pattern.
Brief Title: Sukalmena InAge: Nutritional-culinary Programme to Promote Adherence to a Healthy Dietary Pattern.
Acronym: Sukalmena
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Culinary Center Fundazioa (Other)
Collaborators: University of Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI2021067
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Obesity; Healthy Aging; Cognitive Impairment
Keywords: Mediterranean diet; Culinary intervention; Cooking classes; Nutritional education; Confidence
MeSH Terms: conditions — Obesity; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This study uses a randomized controlled trial design with one-month intervention program and six months of follow-up in order to test the effects of a culinary intervention program to improve cooking and healthy eating behaviour in overweight and obese patients.
  The culinary intervention program will be given over a one-month period, two days a week for four weeks. Participants in the control group (CG) will receive dietary training based on Mediterranean diet at the baseline visit and a leaflet explaining this dietary pattern. The participants assigned to the culinary intervention program will receive the same nutritional recommendations and eight online nutritional and cooking classes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional education group (NEG) (Active Comparator): Participants in the nutritional education group will be given a leaflet with written nutrition educational information to follow a Mediterranean diet. Participants will be encouraged to adhere to this diet for one month. Four visits will be scheduled for participants assigned to this group:
  (1) before randomization (T1); (2) after randomization and before the the beginning of the intervention (T2); and (3) (4) after the intervention (T3)(T4). In all time-points, questionnaires will be registered and at T2 and T4 blood samples will be collected and advanced glycation end-products will be measured.
  Interventions: Behavioral: Mediterranean diet-based nutritional education intervention
- Culinary intervention group (CIG) (Experimental): Participants assigned to the culinary intervention group will receive a written nutrition educational information as well as eight online nutritional and cooking classes during the one-month intervention period. Four visits will be scheduled for participants assigned to this group:
  (1) before randomization (T1); (2) after randomization and before the the beginning of the intervention (T2); and (3) (4) after the intervention (T3)(T4). In all time-points, questionnaires will be registered and at T2 and T4 blood samples will be collected and advanced glycation end-products will be measured.
  Participants will receive 8 culinary workshops between visit 2 and visit 3. In all time-points, questionnaires will be registered and at T2 and T4 blood samples will be collected and advanced glycation end-products will be measured.
  Volunteers will be also contacted by phone after 6 months of the end of the intervention to collect information about food and culinary habits.
  Interventions: Behavioral: Mediterranean diet-based culinary intervention

INTERVENTIONS:
Behavioral: Mediterranean diet-based nutritional education intervention — The patients in the nutritional intervention group will receive dietary advice on how to follow a Mediterranean diet. The dietary recommendations will be given at the beginning of the study by nutritionists using comprehensive written material.
  Arms: Nutritional education group (NEG)
Behavioral: Mediterranean diet-based culinary intervention — The culinary intervention will be developed integrating eight culinary and nutritional workshops that will be given every week, twice per week, during one-month intervention. The duration of each culinary and nutritional workshop will be 1 hour, thus, the program will provide a total of hours of nutritional education and a total of 8 hours of nutritional and cooking training. The courses will take place in a well-equipped kitchen from the Basque Culinary Center and participants will be connected online in order to be able to cook and practice at the same time. All cooking classes will begin with a theoretical introductory part that aim to explain the main take-home messages from the workshop. Subsequently, every class will be characterized by a hands-on part that will include the demonstration and practical preparation of different elaborations based on the use specific cooking techniques and healthy ingredients.
  Arms: Culinary intervention group (CIG)

SUMMARY:
Currently, one of the main health challenges of public health is to improve the quality of life of people with chronic non-communicable diseases, through new strategies that promote healthy eating habits and lifestyles.

Within the new strategies that aim to promote and improve the eating habits of the population, "Sukalmena-InAge" is proposed as a tool for transforming health, where culinary skills and nutritional knowledge converge as a new paradigm to promote health. The merging of culinary knowledge and nutritional education has been coined under the term Culinary Medicine.

The present project is presented as an innovative strategy to improve dietary habits of overweight/obese people. To this end, volunteers will participate in an intervention that will be based on cooking workshops and nutritional education. In this sense, participants will receive different cooking and nutritional education sessions in order to be able to give them resources to cook in an easy, enjoyable and healthy way.

The study will evaluate the effect that this nutritional-culinary intervention programme might exert on health and will compare these results with the effects obtained providing a more traditional nutritional education.

The potential effects will be evaluated through the measurement of specific biochemical parameters related to the most prevalent chronic diseases ( insulin, glucose, total cholesterol, triglycerides, among others). In addition, the measurement of advanced glycation end products (AGEs) in tissue will be carried out. High consumption of AGEs, could induce negative effects on health and has been correlated with the type of food consumed, but also with the culinary techniques used for their preparation.

DETAILED DESCRIPTION:
Lifestyle interventions are nowadays focused on promoting health and preventing chronic diseases. However, when it comes to changing lifestyle habits, and more specifically, dietary habits, the acquisition and maintenance of these modifications over time is often complex due to many factors that may affect.

There is a consensus among health professionals that, based on the available scientific evidence, a diet based on a high consumption of fruit and vegetables is inversely associated with the risk of developing chronic non-communicable diseases and, overall, with lower mortality rates. These protective effects might be in part due to certain nutrients present in the mentioned foods, namely biologically active compounds or bioactive compounds, such as mono- and polyunsaturated fatty acids, fibre, phytochemicals, antioxidant vitamins, minerals, ω-3 fatty acids and plant proteins. These compounds exert antiinflammatory and antioxidant effects, thus, as part of a healthy dietary pattern, they may have the capacity to preserve healthy ageing, for instance, in relation to cognitive status.

Nevertheless, the role of culinary methods from a healthy dietary perspective should not be forgotten. During culinary processes the nutrient content can be modified, contributing not only to the loss or enhancement of beneficial nutrients such as biologically active components (CBAs), but also to the formation of compounds that might be harmful or toxic for the human organism, for example, Advanced Glycation End Products (AGEs).

Taking this into consideration, this study seeks to develop a pilot study to analyse the feasibility and preliminary efficacy of a nutritional-culinary programme aiming to promote long-term healthy ageing in overweight or obese adults. Volunteers participating in the intervention will receive nutritional recommendations based on a healthy dietary pattern such as Mediterranean Diet, together with a culinary training, seeking to empower them in cooking techniques and culinary capacities.

In conclusion, this study aims to evaluate the effectiveness of a nutritional-culinary intervention to produce beneficial effects on health parameters of overweight/obese patients and to compare the results obtained with the health effects obtained through a nutritional intervention without a culinary training.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obesity (BMI between 25 and 35 kg/m2)
* Low score in the screening questionaire "Homecooking Quality Index" (HQI)

Exclusion Criteria:

* Pregnant or lactating women.
* Serious medical condition precluding dietary intervention or limiting survival to less than one year.
* Illicit drug use, chronic alcoholism.
* Participation in any clinical trial with drugs or dietary intervention during the year prior to inclusion.
* Weight loss intervention (surgical treatment, dietary or pharmacological treatment) during the last year
* Difficulty or major drawbacks to change dietary habits and follow Mediterranean diet (allergies, intolerances).

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in adherence to the Mediterranean Diet measured by Mediterranean Diet Adherence Screener (MEDAS) | At baseline, after 4 weeks the beginning of intervention and after 6 months the beginning of intervention
  At baseline, data about adherence to the Mediterranean Diet will be collected by a 14-point Mediterranean Diet Adherence Screener (MEDAS). 4 weeks post-baseline and 6 months post-baseline data from this questionnaire will be also collected. The MEDAS score can range from 0 to 14 and higher scores mean better outcome.
  - Unabbreviated scale title: Mediterranean Diet Adherence Screener
Change in the Frequency of Cooking Habits Questionnaire | At baseline, after 4 weeks the beginning of intervention and after 6 months the beginning of intervention
  At baseline, data about the Frequency of Cooking Habits will be collected by a 24-point questionnaire. 4 weeks post-baseline and 6 months post-baseline, data from this questionnaire will be also collected.
Change in the Confidence towards cooking Questionnaire | At baseline, after 4 weeks the beginning of intervention and after 6 months the beginning of intervention
  At baseline, data about the Confidence towards cooking will be collected by a 18-point questionnaire. 4 weeks post-baseline and 6 months post-baseline data from this questionnaire will be also collected. The Confidence towards cooking questionnaire can range from 18 to 90 and higher scores mean better confidence.
Change in the Attitude towards cooking Questionnaire | At baseline, after 4 weeks the beginning of intervention and after 6 months the beginning of intervention
  At baseline, data about the attitute towards cooking will be collected by a 18-point questionnaire. 4 weeks post-baseline and 6 months post-baseline data from this questionnaire will be also collected. The Attitude towards cooking questionnaire can range from 18 to 90 and higher scores mean better confidence

SECONDARY OUTCOMES:
Change in biochemical parameters (Fasting glucose) | At baseline and after 4 weeks the beginning of intervention
  At baseline blood samples will be collected to measure fasting glucose levels. The second measurement of this parameter will be conducted 4 weeks post-baseline.
Change in biochemical parameters (Fasting insulin) | At baseline and after 4 weeks the beginning of intervention
  At baseline blood samples will be collected to measure fasting insulin level. The second measurement of this parameter will be conducted 4 weeks post-baseline.
Change in biochemical parameters (Fasting total cholesterol) | At baseline and after 4 weeks the beginning of intervention
  At baseline blood samples will be collected to measure fasting total cholesterol levels. The second measurement of this parameter will be conducted 4 weeks post-baseline.
Change in biochemical parameters (Fasting HDL cholesterol) | At baseline and after 4 weeks the beginning of intervention
  At baseline blood samples will be collected to measure fasting HDL cholesterol levels. The second measurement of this parameter will be conducted 4 weeks post-baseline.
Change in biochemical parameters (Fasting LDL cholesterol) | At baseline and after 4 weeks the beginning of intervention
  At baseline blood samples will be collected to measure fasting LDL cholesterol levels. The second measurement of this parameter will be conducted 4 weeks post-baseline.
Change in biochemical parameters (C reactive protein levels) | At baseline and after 4 weeks the beginning of intervention
  At baseline blood samples will be collected to measure fasting C reactive protein levels. The second measurement of this parameter will be conducted 4 weeks post-baseline.
Change in biochemical parameters (TNFalpha) | At baseline and after 4 weeks the beginning of intervention
  At baseline blood samples will be collected to measure TNFalpha levels. The second measurement of this parameter will be conducted 4 weeks post-baseline.
Change in advanced glycation end products (AGEs) level | At baseline and after 4 weeks the beginning of intervention
  At baseline blood samples will be collected for determination of advanced glycation end products levels. 4 weeks post-baseline this determination will be repeated.
Changes in body mass index (BMI) | At baseline and after 4 weeks the beginning of intervention
  BMI will be calculated as body weight (kg) divided by height (m) squared at baseline and 4 weeks post-baseline
Change in fat mass | At baseline and after 4 weeks the beginning of intervention
  At baseline and 4 weeks post-baseline, fat mass will be analyzed by bioimpedance.
Change in fat free mass | At baseline and after 4 weeks the beginning of intervention
  At baseline and 4 weeks post-baseline, fat free mass will be analyzed by bioimpedance.
Changes in hip circumference | At baseline and after 4 weeks the beginning of intervention
  At baseline, hip circumference will be measured with a measuring. 4 weeks post-baseline, the determination of this measurement will be repeated
Changes in waist circumference | At baseline and after 4 weeks the beginning of intervention
  At baseline, waist circumference will be measured with a measuring. 4 weeks post-baseline, the determination of this measurement will be repeated
Change in blood pressure | At baseline and after 4 weeks the beginning of intervention
  At baseline, blood pressure will be measured with a measuring. 4 weeks post-baseline, the determination of this measurement will be repeated
Change in advanced glycation end products (AGEs) in tissue | At baseline and after 4 weeks the beginning of intervention
  At baseline, blood pressure will be measured with a measuring. 4 weeks post-baseline, the determination of this measurement will be repeated.
Change in dietary intake measured by validated Food Frequency Questionnaire (FFQ) | At baseline, after 4 weeks the beginning of intervention and after 6 months the beginning of intervention
  At baseline data about dietary intake will be collected by using a Food Frequency Questionnaire (FFQ) and 4 weeks post-baseline, these data will be collected again. 6 months post-baseline, these data will be also collected. The FFQ is a 136-item questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Usune Etxeberria, PhD, Principal Investigator — BCC Innovation (Basque Culinary Center Fundazioa)
Locations (1):
- Basque Culinary Center Fundazioa, Donostia / San Sebastian, Gipuzkoa, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zaharia OP, Kupriyanova Y, Karusheva Y, Markgraf DF, Kantartzis K, Birkenfeld AL, Trenell M, Sahasranaman A, Cheyette C, Kossler T, Bodis K, Burkart V, Hwang JH, Roden M, Szendroedi J, Pesta DH. Improving insulin sensitivity, liver steatosis and fibrosis in type 2 diabetes by a food-based digital education-assisted lifestyle intervention program: a feasibility study. Eur J Nutr. 2021 Oct;60(7):3811-3818. doi: 10.1007/s00394-021-02521-3. Epub 2021 Apr 11. PMID 33839905
- [Background] Irl B H, Evert A, Fleming A, Gaudiani LM, Guggenmos KJ, Kaufer DI, McGill JB, Verderese CA, Martinez J. Culinary Medicine: Advancing a Framework for Healthier Eating to Improve Chronic Disease Management and Prevention. Clin Ther. 2019 Oct;41(10):2184-2198. doi: 10.1016/j.clinthera.2019.08.009. Epub 2019 Sep 20. PMID 31543284
- [Background] Mills S, White M, Brown H, Wrieden W, Kwasnicka D, Halligan J, Robalino S, Adams J. Health and social determinants and outcomes of home cooking: A systematic review of observational studies. Appetite. 2017 Apr 1;111:116-134. doi: 10.1016/j.appet.2016.12.022. Epub 2016 Dec 23. PMID 28024883
- [Background] Abate G, Marziano M, Rungratanawanich W, Memo M, Uberti D. Nutrition and AGE-ing: Focusing on Alzheimer's Disease. Oxid Med Cell Longev. 2017;2017:7039816. doi: 10.1155/2017/7039816. Epub 2017 Jan 12. PMID 28168012
- [Background] Chou PS, Wu MN, Yang CC, Shen CT, Yang YH. Effect of Advanced Glycation End Products on the Progression of Alzheimer's Disease. J Alzheimers Dis. 2019;72(1):191-197. doi: 10.3233/JAD-190639. PMID 31561370